CLINICAL TRIAL: NCT06168240
Title: THE EFFECT OF MANUAL LYMPHATIC DRAINAGE ON ACUTE AND POST-ACUTE ANKLE SPRAIN IN ATHLETES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sylvia Maher Mohsen Farid Hanna (Other)
Responsible Party: Sponsor-Investigator, Sylvia Maher Mohsen Farid Hanna, master, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/003909
Record Dates: First submitted 2023-11-20; First posted 2023-12-13 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Ankle Sprains
Keywords: Ankle sprain; Athletes; Manual lymphatic drainage
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): will receive Manual lymphatic drainage plus Traditional physical therapy program that will include LASER, cold packs, manual mobilization, and exercise program. Training will applied 3 days a week, for a total of 4 weeks.
  Interventions: Other: Manual lymphatic drainage. will be applied three days per week for four weeks.
- group B (Active Comparator): will receive Traditional physical therapy program only that will include LASER, cold packs, manual mobilization, and exercise program. Training will applied 3 days a week, for a total of 4 weeks.
  Interventions: Other: Manual lymphatic drainage. will be applied three days per week for four weeks.

INTERVENTIONS:
Other: Manual lymphatic drainage. will be applied three days per week for four weeks. — Training will applied 3 days a week, for a total of 4 weeks.
  Other Names: Traditional physical therapy program that will include LASER, cold packs, manual mobilization, and exercise program). will applied three days per week for four weeks.

SUMMARY:
Manual lymphatic drainage techniques (MLDTs) are special techniques in manual therapy used in rehabilitation for treatment of physical dysfunctions and pathologies. Such practices could be done by medical team or clinicians. Theories on MLDTs address functions like stimulating the lymphatic system by increasing lymph circulation, facilitating the removal of waste products from body tissues, reducing edema, and decreasing the responses of sympathetic nervous system while increasing the parasympathetic nervous tone leading to a relaxed body state.

DETAILED DESCRIPTION:
This study will examine the effect of manual lymphatic drainage on pain intensity, ankle swelling, range of motion, static and dynamic functional stability in acute and post-acute ankle sprain in athletes.

Edema treatment includes a variety of techniques; elevation, compression, electrical stimulation, ultrasound, and massage are a few of them. Profound clinical check is required to determine the kind of edema management. However, the effect of these techniques on the lymphatic system and the edema itself is questionable. Manual Lymphatic Drainage mechanism, although still under investigation, is also a valid treatment management that does not cause inflammation, reduces the absorption of waste products and excess fluid and still urges the lymphatic system to work better.

ELIGIBILITY:
Inclusion Criteria:

1. . Basketball Athletes patients diagnosed as acute and post-acute ankle sprain. 2. Patients within 18 and 30 years old. 3. Patients with grade I, II ankle inversion sprain. 4. All participants complains of pain and moderate swelling in the ankle.

Exclusion Criteria:

1. Previous ankle surgery.
2. Serious pathology.
3. History of fractures in the ankle joint.
4. Vascular disorders.
5. Grade III ankle sprain.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
static balance | starting and after 4 weeks
  Flamingo Balance Test to assess static balance
dynamic postural balance | starting and after 4 weeks
  Star Excursion Balance Test to assess dynamic postural balance

SECONDARY OUTCOMES:
Pain intensity | starting and after 4 weeks
  Numeric Pain Rating Scale to assess pain intensity with zero score represents no pain (the better) and ten score represents maximum pain (the worest).
swelling | starting and after 4 weeks
  Figure of Eight with tape measurement by tape measurement to assess swelling in centimeter
range of motion | starting and after 4 weeks
  Goniometer to assess range of motion